CLINICAL TRIAL: NCT03779412
Title: A Randomized Controlled Trial (RCT) Comparing Acceptance and Commitment Therapy (ACT) and Mindfulness-Based Stress Reduction (MBSR) Self-help Books for College Student Mental Health
Brief Title: Self-help Books for Student Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Associate Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9792
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two active self-help interventions for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT self-help book condition (Experimental): Participants in this condition will be assigned to read The Happiness Trap by Harris (2008), a self-help book based on acceptance and commitment therapy.
  Interventions: Behavioral: The Happiness Trap
- MBSR self-help book condition (Active Comparator): Participants in this condition will be assigned to read A Mindfulness-Based Stress Reduction Workbook by Stahl and Goldstein (2010), a self-help book based on Mindfulness-Based Stress Reduction.
  Interventions: Behavioral: A Mindfulness-Based Stress Reduction Workbook

INTERVENTIONS:
Behavioral: The Happiness Trap — Participants assigned to this condition will be asked to read this self-help book over an 8-week period.
  Arms: ACT self-help book condition
Behavioral: A Mindfulness-Based Stress Reduction Workbook — Participants assigned to this condition will be asked to read this self-help book over an 8-week period.
  Arms: MBSR self-help book condition

SUMMARY:
The goal of this study is to compare the efficacy and mechanisms of change of two self-help books for college student mental health in a randomized controlled trial. One book is based on mindfulness-based stress reduction (MBSR), and one is based on acceptance and commitment therapy (ACT).

This study will test the following hypotheses:

1. The ACT and MBSR books will both be feasible and acceptable with college students as evidenced by equivalently high satisfaction and engagement rates.
2. The ACT and MBSR books will be equally effective in improving mental health and well-being among college students.
3. The ACT book will produce larger improvements in valued action, and the MBSR book will produce larger improvements in mindfulness.
4. Valued action will be a stronger predictor of improvements in mental health in the ACT condition and mindfulness will be a stronger predictor of improvements in the mindfulness condition.

DETAILED DESCRIPTION:
The investigators aim to recruit 150 college students for this RCT (75 per treatment condition). This will provide adequate power (0.80) to detect differences between groups of medium effect size (d=0.50). Note that detailed eligibility criteria are listed in the "Eligibility" section. Participants will be recruited via SONA (a participant recruitment system), flyers, online postings, classroom announcements, and through a general online screener for various Utah State University (USU) Contextual Behavioral Science (CBS) Lab studies.

Total study participation will occur over approximately 8 weeks. all study procedures will be completed online, on a computer/mobile phone. After completing informed consent, participants will complete a baseline survey.

At the end of the baseline survey, participants will be randomly assigned to use a book based on ACT (The Happiness Trap) or MBSR (A Mindfulness-Based Stress Reduction Workbook). Participants will be asked not to access other self-help books during the study duration. Participants will be provided with an 8-week reading schedule and a link to the assigned book. Participants will be asked to complete a mid-treatment survey 4 weeks after the beginning of treatment. The mid-treatment survey will include questions about adherence. Participants will be asked to complete a post-treatment survey 8 weeks after the beginning of treatment. This survey will also ask about adherence (reading, use of strategies taught in the book). Researcher contact will involve reminders to complete assessments, basic email assistance in identifying and responding to any barriers to using the self-help book, and twice-weekly reminders of the suggested reading schedule.

After completing the initial assessment participants will be sent a link to The Happiness Trap if they are assigned to the ACT condition, or a link to the Mindfulness-Based Stress Reduction Workbook if they are in the MBSR condition. They will be able to access the book online at any time. Participants will be asked to read assigned chapters on an 8-week schedule.

The Happiness Trap is based on Acceptance and Commitment Therapy, a modern cognitive behavioral therapy that combines acceptance and mindfulness methods with values and behavior change methods. The primary treatment components in The Happiness Trap are psychoeducation of ACT, defusion, acceptance, mindfulness, self-as-context, value, behavioral commitment.

A Mindfulness-Based Stress Reduction Workbook is based on Mindfulness-Based Stress Reduction, a standardized approach to teaching mindfulness, primarily through meditation practices. The primary treatment components in A Mindfulness-Based Stress Reduction Workbook are psychoeducation about mindfulness and mindfulness meditation and various types of mindfulness meditation practice, such as mind-body connection, loving-kindness meditation, interpersonal mindfulness, and the healthy path of mindful eating, exercise, rest, and connection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Enrolled at Utah State University
* Have not participated in other self-help studies run by the USU CBS Lab
* Interested in using self-help book for improving mental health and well-being

Exclusion Criteria:

* Below the age of 18
* Not a student at Utah State University
* Have participated in previous self-help studies run by the CBS Lab
* Not interested in using a self-help book for improving mental health and well-being

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress | Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  Depression, Anxiety and Stress Scale (DASS) : a self-report measure of depression, anxiety, and stress symptoms. Higher scores indicate higher negative emotional states of depression, anxiety, and stress. This measure assesses each of these symptoms as a distinct subscale. Items are rated on a 4-point scale ranging from 0 "did not apply to me at all" to 3 "applied to me very much, or most of the time." Ranges for depression, anxiety, and stress are 0-28, 0-20, and 0-33, respectively.
Change from Baseline Valuing Questionnaire (VQ) at 4 weeks and 8 weeks | Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  A self-report measure of valued action. This is a 10-item measure, and each item is rated on a 7-point scale ranging from 0 "not at all true" to 6 "completely true." The VQ is a new measure, but initial validation results indicate adequate reliability and validity.
Change from Baseline Five Facet Mindfulness Questionnaire (FFMQ) at 4 weeks and 8 weeks. | Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  A self-report measure of five facets of mindfulness: observing, describing, acting with awareness, being nonjudgmental, and nonreactivity. The FFMQ is a 39-item questionnaire, and each FFMQ item is rated on a 5-point scale ranging from 1 ("never or very rarely true") to 5 ("very often or always true"). The FFMQ has been found to be a reliable and valid measure of mindfulness in past research.

SECONDARY OUTCOMES:
Mental Health Continuum - Short Form (MHC-SF) | Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  A self-report measure of positive mental health, composed of three subscales assessing emotional, psychological and social well-being. Items assess theoretically meaningful dimensions of wellbeing including positive affect, satisfaction with life, social integration, social contribution, autonomy, personal growth, purpose in life, and self-acceptance. Items are rated on a 6-point scale ranging from "never" to "every day." The MHC-SF has been found to have adequate reliability and validity in past research.
Counseling Center Assessment of Psychological Symptoms (CCAPS)-Academic Distress Subscale (CCMH, 2012). | Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  The 5-item CCAPS academic distress subscale from the CCAPS-62 will be used to assess academic functioning. Items are rated on a 5-point scale ranging from 0 "not at all like me" to 4 "Extremely like me." The CCAPS has been found to have adequate reliability and validity in past studies with college students.
Acceptance and Action Questionnaire-University Students (AAQ-US). | Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  A self-report measure of psychological inflexibility designed specifically for university students. Items are rated on a 7-point scale ranging from 1 "never true" to 7 "always true." Although this is a new scale, preliminary research supports its reliability and validity.
Cognitive Fusion Questionnaire (CFQ). | Baseline, Baseline, mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  A self-report measure of cognitive fusion, an important process related to mindfulness and ACT. Items are rated on a 7-point scale ranging from 1 "never true" to 7 "always true." Initial validation study found adequate reliability and validity with populations including college students.

OTHER OUTCOMES:
Adherence | Mid-treatment (4 weeks after baseline), and posttreatment (8 weeks after baseline)
  Participants will also be asked to rate their adherence to the exercises in the book on a 7-point scale from "Did all recommended assignments" to "Did no recommended assignments."
Satisfaction with the self-help book | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate 7 items evaluating their satisfaction with the self-help book on a 6-point scale from "Strongly disagree" to "Strongly agree."

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abramowitz JS, Moore EL, Braddock AE, Harrington DL. Self-help cognitive-behavioral therapy with minimal therapist contact for social phobia: a controlled trial. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):98-105. doi: 10.1016/j.jbtep.2008.04.004. Epub 2008 Apr 26. PMID 18514614
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Blanco C, Okuda M, Wright C, Hasin DS, Grant BF, Liu SM, Olfson M. Mental health of college students and their non-college-attending peers: results from the National Epidemiologic Study on Alcohol and Related Conditions. Arch Gen Psychiatry. 2008 Dec;65(12):1429-37. doi: 10.1001/archpsyc.65.12.1429. PMID 19047530
- [Background] Center for Collegiate Mental Health (2012). CCAPS 2012 Technical Manual. University Park, PA
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Harris, R. (2007). The happiness trap: How to stop struggling and start living. Penguin Random House.
- [Background] Hayes, S. C., Strosahl, K. D., & Wilson, K. G. (2011). Acceptance and Commitment Therapy: The process and practice of mindful change. New York: The Guilford Press.
- [Background] Hayes SC, Villatte M, Levin M, Hildebrandt M. Open, aware, and active: contextual approaches as an emerging trend in the behavioral and cognitive therapies. Annu Rev Clin Psychol. 2011;7:141-68. doi: 10.1146/annurev-clinpsy-032210-104449. PMID 21219193
- [Background] Hunt J, Eisenberg D. Mental health problems and help-seeking behavior among college students. J Adolesc Health. 2010 Jan;46(1):3-10. doi: 10.1016/j.jadohealth.2009.08.008. Epub 2009 Oct 20. PMID 20123251
- [Background] Kabat-Zinn J. (1990). Full Catastrophe Living. New York: Delacorte.
- [Background] Keyes CL. Mental illness and/or mental health? Investigating axioms of the complete state model of health. J Consult Clin Psychol. 2005 Jun;73(3):539-48. doi: 10.1037/0022-006X.73.3.539. PMID 15982151
- [Background] Levin ME, Krafft J, Levin C. Does self-help increase rates of help seeking for student mental health problems by minimizing stigma as a barrier? J Am Coll Health. 2018 May-Jun;66(4):302-309. doi: 10.1080/07448481.2018.1440580. Epub 2018 Apr 19. PMID 29447600
- [Background] Levin, M.E., Krafft, J., Pistorello, J. & Seeley, J.R. (In Press). Assessing psychological inflexibility in university students: Development and validation of the acceptance and action questionnaire for university students (AAQ-US). Journal of Contextual Behavioral Science.
- [Background] Levin ME, Pistorello J, Seeley JR, Hayes SC. Feasibility of a prototype web-based acceptance and commitment therapy prevention program for college students. J Am Coll Health. 2014;62(1):20-30. doi: 10.1080/07448481.2013.843533. PMID 24313693
- [Background] Levin, M.E., Stocke, K., Pierce, B. & Levin, C. (2018). Do college students use online self-help? A survey of intentions and use of mental health resources. Journal of College Student Psychotherapy, 32, 181-198.
- [Background] Lovibond, S. H. & Lovibond, P. F. (1995). Manual for the Depression Anxiety Stress Scales, (2nd ed.). Sydney, AU: Psychology Foundation of Australia.
- [Background] McCracken LM, Chilcot J, Norton S. Further development in the assessment of psychological flexibility: a shortened Committed Action Questionnaire (CAQ-8). Eur J Pain. 2015 May;19(5):677-85. doi: 10.1002/ejp.589. Epub 2014 Sep 2. PMID 25181605
- [Background] Rosen, G.M., & Lilienfeld, S.O. (2016). On the failure of psychology to advance self-help: Acceptance and Commitment Therapy (ACT) as a case example. Journal of Contemporary Psychotherapy, 46, 71-77.
- [Background] Sevilla-Llewellyn-Jones J, Santesteban-Echarri O, Pryor I, McGorry P, Alvarez-Jimenez M. Web-Based Mindfulness Interventions for Mental Health Treatment: Systematic Review and Meta-Analysis. JMIR Ment Health. 2018 Sep 25;5(3):e10278. doi: 10.2196/10278. PMID 30274963
- [Background] Smout, M.F., Davies, M., Burns, N., & Christie, A. (2014). Evaluating acceptance and commitment therapy: Development of the valuing questionnaire. Journal of Contextual Behavioral Science, 3, 164-172.
- [Background] Stahl, B. & Goldstein, E. (2010). A Mindfulness-Based Stress Reduction Workbook. New Harbinger Publications